CLINICAL TRIAL: NCT04279795
Title: Study on Detection of 2019 Novel Coronavirus in Multiple Organ System and Its Relationship With Clinical Manifestations in Patients
Brief Title: Detection of 2019 Novel Coronavirus in Multiple Organ System and Its Relationship With Clinical Manifestations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PL11
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Coronavirus
Keywords: 2019 Novel Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Outbreak of 2019 Novel Coronavirus infection quickly spread to the world. Confirmed patients were isolated and treated in our department. 2019 Novel Coronavirus was detected in multiple organ system. Clinical data was recorded to investigate the its relationship with viral detection.

DETAILED DESCRIPTION:
Medical date of suspected patients of 2019 Novel Coronavirus infection, who came to outpatient department of the Third Affiliated Hospital of Sun Yat-sen University, were sent to an expert group if they met the inclusion criteria. The expert group discussed and made a decision if the patient would be admission to isolation unit. Pharyngeal swabs of the patients were obtained and sent to local Center for Disease Control and Prevention (CDC) for detection the 2019 Novel Coronavirus after patients were admission to isolation unit. Diagnosis of 2019 Novel Coronavirus infection was confirmed if the result was positive or excluded if two consecutive results were negative. Patients' demographic data and clinical characteristics were recorded. Clinical characteristics including epidemiological history, past history, personal history, symptoms, signs, blood cells count, biochemical test results, chest computed tomography (CT) images. 2019 Novel Coronavirus RNA was detected in pharyngeal swab, anal swab, urine and blood samples by using quantitative real-time polymerase chain reaction (qPCR). Comprehensive treatments were given to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Epidemiological history including resident of Hubei province, or travel history to Hubei province or exposure to suspected patients in the past two weeks.
2. Symptoms like fever, fatigue, myalgia, headache, cough, sputum production, chest tightness, dyspnea, etc.
3. White blood cells decreased or were normal, or lymphocytes decreased, and chest CT images showed typical findings of viral pneumonia.
4. Detection of 2019 Novel Coronavirus nucleic acid is positive by local Center for Disease Control and Prevention (CDC).

Exclusion Criteria:

1. Patients can not follow-up;
2. Investigator considering inappropriate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed patients of 2019 Novel Coronavirus infection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Positive rate of 2019 Novel Coronavirus RNA | 28 days
  rate of positive results of detection 2019 Novel Coronavirus nucleic acid from urine, blood, anal swabs and pharyngeal swabs samples

SECONDARY OUTCOMES:
Survival rate | 28 days
  If the patient will survive after comprehensive treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China